CLINICAL TRIAL: NCT04914156
Title: The Use of Nutrigenomics in Sports Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Dr Andrea Braakhuis, Academic Director for the Master of Health Sciences in Nutrition & Dietetics, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5000928
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Sport Nutrition; Nutrigenomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised, genetic-based advice for sport performance (Experimental): This group will receive personalised nutrition advice for sports performance based on their genetic test results and tailored to their current dietary intake.
  Interventions: Other: Genetic based dietary advice
- Personalised nutrition advice for sport performance based on population-based evidence (Active Comparator): This group will receive personalised nutrition advice on key nutrients relating to sports performance based on current best practice, population-based sport nutrition guidelines. These will be tailored to their current dietary intake
  Interventions: Other: Personalised population based dietary advice

INTERVENTIONS:
Other: Genetic based dietary advice — Genetic test results for 70 genes relating to nutrition and physical activity will be used in conjunction with participants current dietary intake to create nutrition advice tailored to each individual.
  Arms: Personalised, genetic-based advice for sport performance
Other: Personalised population based dietary advice — Current dietary intake will be compared with current best practice population-based sports nutrition dietary advice to create tailored nutrition advice for each of the participants
  Arms: Personalised nutrition advice for sport performance based on population-based evidence

SUMMARY:
The study's aim is to determine if nutrigenomics-based dietary advice is a greater motivator for dietary change amongst an athlete population. Specifically, the investigators will be examining whether nutrigenomics-based personalized dietary advice results in greater changes in dietary intake and body composition amongst athletes compared to personalised population-based sports nutrition advice. It is hypothesized that the Nutrigenomics in Sports Nutrition group would engage in greater dietary changes and better adhere to the dietary advice compared to the standard advice group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Competes in representative sports team
* Has access to the internet and smart phone device
* Able to speak English

Exclusion Criteria:

* N/A

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Changes in dietary intake from baseline | 8 weeks
  We will assess dietary intake for energy intake, carbohydrates, protein, fat, sodium, caffeine, glycemic index, iron, Vitamin A, Vitamin B12, Vitamin C, Vitamin D, Vitamin E, Folate and Calcium using a 3 day food record conducted at baseline using Easy Diet Diary phone application. A second 3 day food record will be conducted post intervention period to examine any changes in dietary habits.

SECONDARY OUTCOMES:
Changes in body composition from baseline | 8 weeks
  At baseline, participants will indicate body composition goals and baseline body composition measurements will be taken using International Society for Advancement of Kinanthropometry accredited guidelines. Repeated body composition measurements will be taken post intervention to examine in any changes in body composition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Auckland, Auckland, New Zealand